CLINICAL TRIAL: NCT06036992
Title: Study and Management of Cystic Complications in Autosomal Dominant Polycystic Kidney Disease
Acronym: COMPLIK
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC22.0232 - COMPLIK
Record Dates: First submitted 2023-06-26; First posted 2023-09-14 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Polycystic Kidney Diseases
MeSH Terms: conditions — Polycystic Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Autosomal dominant polycystic kidney disease is characterised by the development of renal and hepatic cysts. While the main complication is chronic end-stage renal failure, specific cyst-related complications are common: intracystic haemorrhage, renal or hepatic cyst infections, cyst-related mechanical complications and lithiasis. To date, there is no reliable epidemiological data on the frequency and clinical impact of these complications. Diagnosis of these complications is often complicated, and their management has not been codified. The latest international recommendations (KDIGO) provide only low-level recommendations. For the most complex cases (recurrent cystic infections, resistant pain, mechanical complications and malnutrition, need for pre-transplant nephrectomy, etc.), practitioners are often at a loss and management varies greatly from one centre to another.

DETAILED DESCRIPTION:
Autosomal dominant polycystic kidney disease is characterised by the development of renal and hepatic cysts. While the main complication is chronic end-stage renal failure, specific cyst-related complications are common: intracystic haemorrhage, renal or hepatic cyst infections, cyst-related mechanical complications and lithiasis. To date, there is no reliable epidemiological data on the frequency and clinical impact of these complications. Diagnosis of these complications is often complicated, and their management has not been codified. The latest international recommendations (KDIGO) provide only low-level recommendations. For the most complex cases (recurrent cystic infections, resistant pain, mechanical complications and malnutrition, need for pre-transplant nephrectomy, etc.), practitioners are often at a loss and management varies greatly from one centre to another.

ELIGIBILITY:
Inclusion Criteria:

* Patient with autosomal dominant polycystic kidney disease (APKD) participating in the Genkyst study
* Patient with at least one cystic complication. The cystic complications retained are the following:

  * Acute or chronic cyst-related pain requiring analgesic treatments
  * Cyst infection
  * Intracystic haemorrhage
  * Urinary lithiasis
  * Functional complaints related to the cystic mass: digestive disorders with eating disorders, undernutrition, diaphragmatic compression phenomena, portal hypertension, umbilical or linea alba hernias, ventrations
  * Need for a cystic reduction procedure: puncture, marsupialization, open surgery (including preparation for grafting)

Exclusion Criteria:

* Patients who have expressed their opposition to taking part in the study
* Patient under legal protection (guardianship, curatorship, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with autosomal dominant polycystic kidney disease included in Genkyst who present at least one cystic complication.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
To improve knowledge of the epidemiology of cystic complications within the Genkyst network | 12 months
  number of cases of cystic complications per year per complication

SECONDARY OUTCOMES:
Creation of a specific multidisciplinary consultation meeting | 12 months
  Meetings and exchanges between different health professionals: interventional radiologists, surgeons, infectiologists, hepatologists, pain specialists and nephrologists to discuss the best possible management for patients with complex cystic complications.
Creation of an image bank | 12 months
  consulting images to recalculate and improve diagnostic scores
Creation of a group of control patients | 12 months
  the change from baseline in quality of life scores at 1 year.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.